CLINICAL TRIAL: NCT03533257
Title: Phase II Study to Assess the Safety, Tolerability, and Target Engagement of AMX0035, a Fixed Combination of Sodium Phenylbutyrate and Tauroursodeoxycholic Acid for the Treatment of Alzheimer's Disease
Brief Title: Study to Assess the Safety and Biological Activity of AMX0035 for the Treatment of Alzheimer's Disease
Acronym: PEGASUS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amylyx Pharmaceuticals Inc. (Industry)
Collaborators: Alzheimer's Drug Discovery Foundation (Other); Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMX-8000
Record Dates: First submitted 2018-04-30; First posted 2018-05-23 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — sodium phenylbutyrate and taurursodiol; 4-phenylbutyric acid; ursodoxicoltaurine

STUDY DESIGN:
Intervention Model Description: Placebo-Controlled, Double-Blind, Parallel-Group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (AMX0035) (Active Comparator): AMX0035 twice daily--a combination of Sodium Phenylbutyrate (3g) and Taurursodiol (1g)
  Interventions: Drug: AMX0035
- Placebo (Placebo Comparator): Taste-matched Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMX0035 — Combination Therapy of PB and TURSO
  Other Names: Sodium Phenylbutyrate (PB) and Taurursodiol (TURSO; also known as Tauroursodeoxycholic Acid [TUDCA])
  Arms: Active (AMX0035)
Drug: Placebo — Placebo
  Other Names: Comparator
  Arms: Placebo

SUMMARY:
The study is a 24-week, randomized, double-blind, multi-site, placebo-controlled study in participants with mild cognitive impairment (MCI) or early dementia due to Alzheimer's disease (AD).

DETAILED DESCRIPTION:
The study is a 24-week, randomized, double-blind, multi-site, placebo-controlled study in participants with mild cognitive impairment (MCI) or early dementia due to Alzheimer's disease (AD). The study is designed to evaluate the safety, tolerability, drug target engagement and neurobiological effects of treatment with AMX0035 over 24 weeks. The study is designed to yield deep phenotyping insight for the purposes of demonstrating the effects of AMX0035 on mechanistic targets of engagement and disease biology. The study will evaluate diverse disease-relevant markers and produce an informative dataset that will allow for evaluation and correlation of imaging-based markers, neurobiological changes, functional measures, and cognitive outcomes. Participants receive orally administered study drug twice daily for a treatment duration of approximately 24 weeks and attend clinic visits at Screening, Baseline, Week 6, Week 12, Week 18, and Week 24.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 55-89, inclusive, male or female
2. Diagnosis of "Probable Alzheimer's Disease" or Mild Cognitive Impairment (amnestic or amnestic plus other) with biomarkers that suggest intermediate or high likelihood that the syndrome is due to AD, according to 2011 NIA-AA Workgroup criteria
3. MoCA score >/=8
4. Able to read and write in English sufficiently to complete all study procedures
5. Geriatric Depression Scale <7
6. Willing and able to complete all assessments and study procedures
7. Not pregnant, lactating or of child-bearing potential (women must be >2 years post-menopausal or surgically sterile)
8. Study partner with at least two days per week with contact with patient willing to accompany patient to visits and complete partner study forms
9. No known hypersensitivity to TURSO or Phenylbutyrate
10. If on cholinesterase inhibitor and/or memantine, treatment must have started for no less than 3 months (84 days) prior to baseline and the dosing regimen must have remained stable for 6 weeks (42 days) prior to baseline. The Investigator anticipated that the dosing regimen at baseline would remain unchanged throughout participation in the study.

Exclusion Criteria:

1. Any CNS disease other than suspected AD, such as clinical stroke, brain tumor, normal pressure hydrocephalus, multiple sclerosis, significant head trauma with persistent neurological cognitive deficits or complaints, Parkinson's disease, frontotemporal dementia, or other neurodegenerative diseases
2. Abnormal liver function defined as AST and/or ALT > 3 times the upper limit of normal
3. Renal insufficiency as defined by a serum creatinine > 1.5 times the upper limit of normal
4. Recent (less than 1 year) cholecystectomy or the presence of post-cholecystectomy syndrome or biliary obstruction
5. Clinically significant unstable medical condition (other than AD) that in the Site Investigator opinion would pose a risk to the participant if they were to participate in the study
6. Any contraindication to undergo MRI studies such as:

   1. History of a cardiac pacemaker or pacemaker wires
   2. Metallic particles in the body
   3. Vascular clips in the head
   4. Prosthetic heart valves
   5. Severe claustrophobia impeding ability to participate in an imaging study, or

   MRI findings that show one or more of the following:
   1. More than 4 incidental microhemorrhages
   2. Incidental lacunar infarct with attributable signs or symptoms and with history of stroke
   3. Incidental meningiomas with attributable signs or symptoms
   4. Newly recognized meningioma
7. Major active or chronic psychiatric illness (e.g. depression, bipolar disorder, obsessive compulsive disorder, schizophrenia) that is not stable or well controlled within the previous year prior to baseline
8. Any significant neurodevelopmental disability
9. Current suicidal ideation or history of suicide attempt within 5 years of baseline or significant change from the screening and baseline C-SSRS at the discretion of the Site Investigator
10. History of alcohol or other substance abuse or dependence within the past 2 years
11. Any significant systemic illness or medical condition that could affect safety or compliance with study at the discretion of the Site Investigator
12. Laboratory abnormalities in B12, TSH, or other common laboratory parameters that might contribute to cognitive dysfunction
13. Current use of medications with psychoactive properties that may deleteriously affect cognition (e.g., anticholinergics, centrally-acting antihistamines, antipsychotics, sedative hypnotics, anxiolytics)
14. Use of any investigational therapy being used or evaluated for the treatment of AD is prohibited beginning 3 months (90 days) prior to the Baseline Visit and throughout the study.
15. Use of other investigational agents 1 month (28 days) prior to the Baseline Visit and for the duration of the trial.

Ages: 55 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Yeramian, MD, Study Director — Amylyx Pharmaceuticals Inc.
Locations (11):
- United States (11):
  - Clinical Neuroscience Solutions, Inc. - Jacksonville, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc. - Orlando, Orlando, Florida
  - International Medical Investigational Centers (IMIC), Palmetto Bay, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Rowan University School of Osteopathic Medicine, Stratford, New Jersey
  - Mount Sinai Alzheimer's Disease Research Center, New York, New York
  - Columbia University, New York, New York
  - Hospital of the University of Pennsylvania, Penn Memory Center, Philadelphia, Pennsylvania
  - Genesis NeuroScience Clinic, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arnold SE, Hendrix S, Nicodemus-Johnson J, Knowlton N, Williams VJ, Burns JM, Crane M, McManus AJ, Vaishnavi SN, Arvanitakis Z, Neugroschl J, Bell K, Trombetta BA, Carlyle BC, Kivisakk P, Dodge HH, Tanzi RE, Yeramian PD, Leslie K. Biological effects of sodium phenylbutyrate and taurursodiol in Alzheimer's disease. Alzheimers Dement (N Y). 2024 Aug 9;10(3):e12487. doi: 10.1002/trc2.12487. eCollection 2024 Jul-Sep. PMID 39131742
- [Derived] Wen ZQ, Lin J, Xie WQ, Shan YH, Zhen GH, Li YS. Insights into the underlying pathogenesis and therapeutic potential of endoplasmic reticulum stress in degenerative musculoskeletal diseases. Mil Med Res. 2023 Nov 9;10(1):54. doi: 10.1186/s40779-023-00485-5. PMID 37941072
- See also: "Biological effects of sodium phenylbutyrate and taurursodiol in Alzheimer's disease" — https://pubmed.ncbi.nlm.nih.gov/39131742/

RESULTS

PARTICIPANT FLOW:
Groups:
- Active (AMX0035): AMX0035 twice daily--a combination of Sodium Phenylbutyrate (PB) and Taurursodiol (TURSO)
Period: Overall Study
Arm/Group | Active (AMX0035) | Placebo
Started | 51 | 44
Completed | 41 | 42
Not Completed | 10 | 2
Not completed — Adverse Event | 4 | 2
Not completed — Enrolled in other study, terminated by Sponsor, other | 6 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Active (AMX0035) | Placebo | Total
Number analyzed (Participants) | 51 | 44 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.7 (7.69) | 70.7 (7.30) | 70.7 (7.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 19 | 43
  Male | 27 | 25 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 49 | 43 | 92
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 51 | 44 | 95
ApoE4 Gene Group 1 [Count of Participants; unit: Participants]
  Carrier | 37 | 27 | 64
  Non-carrier | 11 | 17 | 28
  Not reported | 3 | 0 | 3
ApeE4 Gene Group 2 [Count of Participants; unit: Participants]
  1 allele | 29 | 18 | 47
  2 alleles | 8 | 9 | 17
  Non-carrier | 11 | 17 | 28
  Not reported | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Event (TEAEs)
Description: Comparison between the AMX0035 Group and Placebo of the number of participants with TEAEs
Time Frame: From first dose to 24 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Active (AMX0035) | Placebo
Number analyzed (Participants) | 51 | 44
Participants | 34 | 26

2. Primary Outcome: Effect of Treatment on a Global Composite Statistical Test of Cognition, Function, and Neuroanatomy (GST)
Description: Change from Baseline in GST (global statistical test combining three measures relevant to disease trajectory (cognition [MADCOMS: Mild/Moderate Alzheimer's Disease Composite Score], function [FAQ: Functional Activities Questionnaire], and total hippocampal volume on magnetic resonance imaging)) for AMX0035 relative to placebo. For MADCOMS and FAQ, a higher score indicates a worse outcome. A larger hippocampal volume is better, so it was reversed before being normalized. Each of the three were normalized against respective baseline means and standard deviations. The mean of the three normalized scores is the final GST. A higher GST score indicates a worse outcome. Standard deviations above the mean are worse; standard deviations below the mean are better.
  The expected value of the GST at baseline is 0 because it is the mean of three z-scores whose expected values at baseline are 0. AD is multifaceted and the GST was designed to be sensitive to changes in multiple dimensions.
Time Frame: 24 weeks
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active (AMX0035) | Placebo
Number analyzed (Participants) | 51 | 44
score on a scale | 0.24 (0.049) | 0.17 (0.052)
Statistical Analysis 1: Comparison: Active (AMX0035) vs Placebo; Test type: Superiority; p = 0.3654, Mixed Models Analysis; The analysis assessed the difference in estimated change-from-baseline values at the 24-week model estimate using LS means estimates from the MMRM

3. Secondary Outcome: Effect of Treatment on Cognition
Description: Impact of AMX0035 on clinical symptoms as measured by Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog). Scoring is in the range of 0 to 90 with a higher score indicating greater cognitive impairment.
Time Frame: 24 weeks
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active (AMX0035) | Placebo
Number analyzed (Participants) | 51 | 44
score on a scale | 2.26 (1.402) | 1.52 (1.496)
Statistical Analysis 1: Comparison: Active (AMX0035) vs Placebo; Test type: Superiority; p = 0.6698, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

4. Secondary Outcome: Effect of Treatment on Functioning
Description: Impact of AMX0035 on Functional Activities Questionnaire (FAQ) scores. FAQ total score can range from 0 to 30, with higher scores indicating less functional independence.
Time Frame: 24 weeks
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active (AMX0035) | Placebo
Number analyzed (Participants) | 51 | 44
score on a scale | 2.61 (0.790) | 1.59 (0.845)
Statistical Analysis 1: Comparison: Active (AMX0035) vs Placebo; Test type: Superiority; p = 0.3086, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

5. Secondary Outcome: Effect of Treatment on Dementia Severity
Description: Impact of AMX0035 on Dementia Severity Rating Scale (DSRS) scores. Total score can range from 0 to 54, with higher scores indicating greater severity of dementia.
Time Frame: 24 weeks
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active (AMX0035) | Placebo
Number analyzed (Participants) | 51 | 44
score on a scale | 2.34 (0.595) | 1.81 (0.636)
Statistical Analysis 1: Comparison: Active (AMX0035) vs Placebo; Test type: Superiority; p = 0.5552, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

6. Secondary Outcome: Effect of Treatment on Cognitive Impairment
Description: Impact of AMX0035 on the Montreal Cognitive Assessment (MoCA) scores. MoCA scores can range from 0 to 30, with lower scores indicating greater cognitive impairment.
Time Frame: 24 weeks
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active (AMX0035) | Placebo
Number analyzed (Participants) | 51 | 44
score on a scale | -2.18 (0.483) | -0.70 (0.512)
Statistical Analysis 1: Comparison: Active (AMX0035) vs Placebo; Test type: Superiority; p = 0.0361, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

7. Secondary Outcome: Effect of Treatment on Neuropsychiatric Symptoms
Description: Impact of AMX0035 on neuropsychiatric symptoms as assessed by the Neuropsychiatric Inventory (NPI). The total score ranges from 0 to 36, with higher scores indicating a greater severity of symptoms.
Time Frame: 24 weeks
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active (AMX0035) | Placebo
Number analyzed (Participants) | 51 | 44
score on a scale | 0.15 (0.490) | -0.46 (0.526)
Statistical Analysis 1: Comparison: Active (AMX0035) vs Placebo; Test type: Superiority; p = 0.3585, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

8. Secondary Outcome: Regional Brain Volume
Description: Impact of AMX0035 on levels of hippocampal atrophy, as assessed by volumetric Magnetic Resonance Imaging (vMRI)
Time Frame: 24 weeks
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | Active (AMX0035) | Placebo
Number analyzed (Participants) | 51 | 44
mm^3 | -75.18 (25.429) | -70.78 (23.308)
Statistical Analysis 1: Comparison: Active (AMX0035) vs Placebo; Test type: Superiority; p = 0.8996, Mixed Models Analysis; [statistical method as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: 24 weeks
Groups:
- Active (AMX0035): AMX0035--a combination of Sodium Phenylbutyrate (PB) and Taurursodiol (TURSO)
Arm/Group | Active (AMX0035) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/44
Serious Adverse Events (participants affected / at risk) | 3/51 | 1/44
Other Adverse Events (participants affected / at risk) | 12/51 | 6/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (AMX0035) (N=51) | Placebo (N=44)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active (AMX0035) (N=51) | Placebo (N=44)
Diarrhoea (Gastrointestinal disorders) | 8 | 3
Headache (Nervous system disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT03533257/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT03533257/SAP_001.pdf